CLINICAL TRIAL: NCT02809781
Title: Phase III Study of Human Bone Marrow-Derived Mesenchymal Stem Cells to Treat AS
Brief Title: A Pilot Study of MSCs Iufusion and Etanercept to Treat Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shen Huiyong, Director of Orthopedics, Sun Yat-sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-81332612
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Spondylitis; Spondylitis, Ankylosing; Ankylosis; Arthritis; Spondylarthritis; Spondylarthropathies; Spinal Diseases; Musculoskeletal Diseases; Bone Diseases
Keywords: ankylosing spondylitis; mesenchymal stem cell; etanercept
MeSH Terms: conditions — Spondylitis; Spondylitis, Ankylosing; Ankylosis; Arthritis; Spondylarthritis; Spondylarthropathies; Spinal Diseases; Musculoskeletal Diseases; Bone Diseases | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous infusion of MSCs (Experimental): Human bone marrow-derived MSCs at a dose of 1.0E+6 MSC/kg, receive infusion per week in the first 4 weeks and every two weeks in the second 8 weeks. total for 12 weeks.
  Interventions: Biological: Intravenous infusion of MSCs
- Etanercept (Active Comparator): 50mg,hypodermic injection,once per week, for 12 weeks
  Interventions: Drug: Etanercept

INTERVENTIONS:
Biological: Intravenous infusion of MSCs — Intravenous infusion of MSCs:Human bone marrow-derived MSCs 1.0E+6 MSC/kg, IV drop
  Arms: Intravenous infusion of MSCs
Drug: Etanercept — 50mg,hypodermic injection,once per week, for 12 weeks
  Other Names: TNF alpha receptor inhibitor
  Arms: Etanercept

SUMMARY:
The purpose of this study is to evaluate the safety and clinical effect of mesenchymal stem cells (MSCs) derived from human bone marrow at a dose of 1.0E+6 MSC/kg in subject for the therapy of Ankylosing spondylitis (AS) and to compare the efficacy of MSCs and Etanercept to treat this disease.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic, progressive inflammatory rheumatic disease involving primarily the sacroiliac joints and the axial skeleton. The main clinical features are back pain and progressive stiffness of the spine. Oligoarthritis of the hips and shoulders, enthesopathy, and anterior uveitis are common, and involvement of the heart and lungs is rare. The current understanding of the pathogenesis of this disorder is limited.It mainly about to hereditary susceptibility (eg HLA-B27),infection and autoimmunity.

Although traditional drugs, such as Nonsteroidal antiinflammatory drugs (NSAIDs) disease-modifying antirheumatic drugs (DMARDs such as methotrexate, salicylazosulfapyridine OR thalidomide) and steroids have been used in the treatment of AS, however, many studies have indicated that the overall response to these drugs is not satisfied. Addition, the severe side effects of these drugs have also been observed. The management of AS patients therefore remains unsatisfactory and targeted therapies are needed. Although the application of TNF alpha receptor inhibitor (such as Etanercept) has got the success in the early treatment of ankylosing spondylitis, the tolerance to this biological agent make the therapy to this disease rather difficult. Recently, owning to its immunoregulatory, immunosuppressive, stimulating hematopoiesis and tissue repairing properties, the infusion of human MSCs isolated from human bone marrow have been a promising and effective treatment to AS patients. This study will evaluate the safety and effectiveness of MSC transplantation in the AS patients and compare the efficiency with the Etanercept to treat AS patients.

This study will last 2 to 3 years. Participants will be randomly assigned to receive either MSC transplant therapy (experimental group) or Etanercept therapy (control group). Patients will undergo MSC transplant at the start of the study on Day 0. The experimental group will receive infusion per week in the first 4 weeks and every two weeks in the second 8 weeks, totally for 12 weeks. After 3 months, patients will receive the second MSC transplantation. After 12 weeks (Phase I) and 48 weeks (Phase II) from the first transplantation, patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The male or female patient aged 18 to 45 years;
2. Fulfill 1984 modified NewYork classification criteria for AS;
3. The score of the Bath AS Disease Activity Index (BASDAI)≥40 on (0-100) despite optimal non-steroidal anti-inflammatory drug (NSAID) treatment.
4. Before each experiment, patients subscribe voluntarily to the agreement approved by Ethics Committees and sign the date.

Exclusion Criteria:

1. The patient diagnosed in doubt;
2. Completely stiff spine
3. Received spinal or joint surgery within 2 months
4. Received anti-TNF therapy within 3 months
5. pregnant or suckling period female patients;
6. Patients with the Medical or mentally imbalance charged by researchers. patients associated cardiovascular, cerebrovascular, liver,renal and hematological system diseases or mental disease;
7. Patients could not accept the research or could not cooperate well. Patients with other sever diseases at the same time, such as abnormality of joints, other seronegative spondyloarthropathy, or other Rheumatic Diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The Assessment of Spondyloarthritis International Society (ASAS)20 response | 48 weeks
  ASAS measures symptomatic improvement in AS patients.ASAS=4 domains:patient global assessment of disease activity,pain,function,inflammation.ASAS 20=20% improvement(vs.baseline)and an absolute change≥1 units on a 0-10 scale(0=no disease activity;10=high disease activity)for ≥3 domains,and no worsening in remaining domain.

SECONDARY OUTCOMES:
BASDAI score comparing to baseline | 48 weeks
BASFI score comparing to baseline | 48 weeks
  the Bath Ankylosing Spondylitis Functional Index
Imageology | 48 weeks
  The bone marrow of the whole spine (from C2 to S1) can be detected by Magnetic resonance imaging (MRI) scan. The MRI sequence included a T1-weighted turbo spin-echo (TSE) sequence and a fat-saturated short tau inversion recovery (STIR) sequence.
  MR images were first analyzed using the ASspiMRI-a scoring system , which is based on grading disease activity on a scale of 0 to 6. In addition to the ASspiMRI-a scoring system, the inflammation area and average intensityof each inflammatory site were calculated. The background value (BV) was obtained by taking 10 normal sites of the vertebral body of 1 layer and calculating the average. The inflammation extent of each inflammatory site was calculated by the formula:
  value of inflammation area (VIA) × [value of average intensity (VAI) - BV]. The summation of the inflammation extent of all inflammatory sites in all scanning layers was defined as the total inflammation extent (TIE) of each patient.
C-reactive protein (CRP) | 12 weeks
Erythrocyte sedimentation rate (ESR) | 12 weeks
Tumor necrosis factor alpha (TNF-α) | 12 weeks
Interleukin 6 (IL-6) | 12 weeks
Interleukin 17 (IL-17) | 12 weeks

OTHER OUTCOMES:
Percentage of systemic T cell population | 12 weeks
Side effects | 48 weeks
  These parameters monitored throughout the trial included body temperature, pulse rate, respiration rate, blood pressure, complete blood count (CBC), routine urine and stool testing, blood creatinine, alanine transaminase, and aspartate transaminase levels, anti-nuclear antibody testing, electrocardiogram, and chest radiographs. These data were obtained by skilled allied health professionals strictly according to the international standardized procedure when patients were enrolled in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Huiyong, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
It all depends on the whole process of the study.